CLINICAL TRIAL: NCT06453603
Title: Efficacy of Platelet-rich Plasma Injection Compare With Corticosteroid in Pes Anserinus Pain Syndrome, Randomized Controlled Trial Study
Brief Title: Efficacy of Platelet-rich Plasma Injection Compare With Corticosteroid in Pes Anserinus Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Thaned Ekthanaporn, Doctor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pending 00
Record Dates: First submitted 2024-05-23; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pes Anserine Bursitis; Steroid Injection; PRP Injection
Keywords: Pes Anserine Bursitis; Steroid Injection; PRP injection
MeSH Terms: conditions — Bursitis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP injection (Experimental): receive pes anserinus PRP injection
  Interventions: Drug: PRP injection
- Corticosteroid injection (Active Comparator): receive pes anserinus corticosteroid injection
  Interventions: Drug: corticosteroid injection

INTERVENTIONS:
Drug: PRP injection — Receive pes anserinus PRP injection
  Arms: PRP injection
Drug: corticosteroid injection — Receive pes anserinus corticosteroid injection
  Arms: Corticosteroid injection

SUMMARY:
The goal of this research is to study the efficacy of treatment between PRP injection and corticosteroid injection in patients with pes anserinus bursitis. The research question is whether PRP can reduce pain more effectively than corticosteroids.

The study is divided into two groups: one group receiving PRP injections and the second group receiving corticosteroid injections. Treatment outcomes will be monitored at four time points: baseline, 4 weeks, 12 weeks, and 24 weeks. The outcomes will be measured using the VAS and WOMAC scores.

DETAILED DESCRIPTION:
Randomization of patient with pes anserinus bursitis at opd od ramathibodi hospital.

Objective : to study the efficacy of treatment between PRP injection and corticosteroid injection in patients with pes anserinus bursitis

Medhods :

A randomized controlled trial , Single blinded Participants : Patients with pes anserinus bursitis Randomization : Randomization will be performed using the software STATA 16.0 (StataCorp, College Station, Texas, USA). A various blocked randomization method

Interventions and control :

* Experimental groups : PRP injection 4 ml
* Control groups : Steroid injection , Triamcinolone acetonide(40mg/ml) 1 ml + 1%Lidocaine without adrenaline 3 ml = 4ml By Orthopedic surgeon with ultrasound guide.

Allocation and concealment :

A central randomization service will prepare sealed envelopes containing the assigned treatment for each patient.

The envelopes will be kept in secure location until Break the concealment at outpatient orthopedics department , Ramathibodi hospital

Blinding :

Randomized controlled trial study, Single blinded The assessor who will be follow up the patients, will be blinded to the group assignments.

Outcome measures:

Visual Analogue Scale (VAS) , Womac scores

Follow up:

at 4 weeks, 12 weeks, and 24 weeks after injection.

Statistic analysis:

STATA 16.0, StataCorp, College Station, Texas, USA Analysis Demographic data : mean, SD Mean difference in patient-relevant outcomes : Independent T- test

ELIGIBILITY:
Inclusion Criteria

* Over 18 years old
* Patients diagnosed with Pes Anserine Pain Syndrome
* Patients willing to participate in the research project by signing a consent form

Exclusion Criteria:

* Patients with a localized knee infection or a disseminated infection within the past 3 months
* Patients with thyroid disorders, rheumatoid arthritis, or other types of knee arthritis
* Patients with abnormal blood coagulation or thrombocytopenia
* Patients who are pregnant
* Patients with any type of cancer
* Patients who cannot follow up with treatment until the end of the project
* Patients who are unwilling to participate in the project or wish to withdraw from the research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 6 months
  Pain relief outcome : Visual analogue scale (VAS) scale 0(minimum pain) to 10(maximum pain)

SECONDARY OUTCOMES:
WOMAC score | 6 months
  Functional outcomes : The Western Ontario and McMaster Universities Arthritis Index(WOMAC) version 3.01 Thai version

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuptniratsaikul V, Rattanachaiyanont M. Validation of a modified Thai version of the Western Ontario and McMaster (WOMAC) osteoarthritis index for knee osteoarthritis. Clin Rheumatol. 2007 Oct;26(10):1641-5. doi: 10.1007/s10067-007-0560-y. Epub 2007 Feb 20. PMID 17310271
- [Result] Yoon HS, Kim SE, Suh YR, Seo YI, Kim HA. Correlation between ultrasonographic findings and the response to corticosteroid injection in pes anserinus tendinobursitis syndrome in knee osteoarthritis patients. J Korean Med Sci. 2005 Feb;20(1):109-12. doi: 10.3346/jkms.2005.20.1.109. PMID 15716614
- [Result] Saltzman BM, Leroux T, Meyer MA, Basques BA, Chahal J, Bach BR Jr, Yanke AB, Cole BJ. The Therapeutic Effect of Intra-articular Normal Saline Injections for Knee Osteoarthritis: A Meta-analysis of Evidence Level 1 Studies. Am J Sports Med. 2017 Sep;45(11):2647-2653. doi: 10.1177/0363546516680607. Epub 2016 Dec 27. PMID 28027657
- [Result] Subotnick SI, Sisney P. Treatment of Achilles tendinopathy in the athlete. J Am Podiatr Med Assoc. 1986 Oct;76(10):552-7. doi: 10.7547/87507315-76-10-552. No abstract available. PMID 3772761
- [Result] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Result] Wong MW, Tang YY, Lee SK, Fu BS, Chan BP, Chan CK. Effect of dexamethasone on cultured human tenocytes and its reversibility by platelet-derived growth factor. J Bone Joint Surg Am. 2003 Oct;85(10):1914-20. doi: 10.2106/00004623-200310000-00008. PMID 14563798
- [Result] Liu D, Ahmet A, Ward L, Krishnamoorthy P, Mandelcorn ED, Leigh R, Brown JP, Cohen A, Kim H. A practical guide to the monitoring and management of the complications of systemic corticosteroid therapy. Allergy Asthma Clin Immunol. 2013 Aug 15;9(1):30. doi: 10.1186/1710-1492-9-30. PMID 23947590
- [Result] Han SH, An HJ, Song JY, Shin DE, Kwon YD, Shim JS, Lee SC. Effects of corticosteroid on the expressions of neuropeptide and cytokine mRNA and on tenocyte viability in lateral epicondylitis. J Inflamm (Lond). 2012 Oct 30;9(1):40. doi: 10.1186/1476-9255-9-40. PMID 23107345
- [Result] Carofino B, Chowaniec DM, McCarthy MB, Bradley JP, Delaronde S, Beitzel K, Cote MP, Arciero RA, Mazzocca AD. Corticosteroids and local anesthetics decrease positive effects of platelet-rich plasma: an in vitro study on human tendon cells. Arthroscopy. 2012 May;28(5):711-9. doi: 10.1016/j.arthro.2011.09.013. Epub 2012 Jan 21. PMID 22264830
- [Result] Ahmad Z, Siddiqui N, Malik SS, Abdus-Samee M, Tytherleigh-Strong G, Rushton N. Lateral epicondylitis: a review of pathology and management. Bone Joint J. 2013 Sep;95-B(9):1158-64. doi: 10.1302/0301-620X.95B9.29285. PMID 23997125
- [Result] Everts P, Onishi K, Jayaram P, Lana JF, Mautner K. Platelet-Rich Plasma: New Performance Understandings and Therapeutic Considerations in 2020. Int J Mol Sci. 2020 Oct 21;21(20):7794. doi: 10.3390/ijms21207794. PMID 33096812
- [Result] Uysal F, Akbal A, Gokmen F, Adam G, Resorlu M. Prevalence of pes anserine bursitis in symptomatic osteoarthritis patients: an ultrasonographic prospective study. Clin Rheumatol. 2015 Mar;34(3):529-33. doi: 10.1007/s10067-014-2653-8. Epub 2014 May 6. PMID 24797774
- [Result] Kemp JA, Olson MA, Tao MA, Burcal CJ. Platelet-Rich Plasma versus Corticosteroid Injection for the Treatment of Lateral Epicondylitis: A Systematic Review of Systematic Reviews. Int J Sports Phys Ther. 2021 Jun 1;16(3):597-605. doi: 10.26603/001c.24148. PMID 34123513
- [Result] Gautam VK, Verma S, Batra S, Bhatnagar N, Arora S. Platelet-rich plasma versus corticosteroid injection for recalcitrant lateral epicondylitis: clinical and ultrasonographic evaluation. J Orthop Surg (Hong Kong). 2015 Apr;23(1):1-5. doi: 10.1177/230949901502300101. PMID 25920633
- [Result] Ben-Nafa W, Munro W. The effect of corticosteroid versus platelet-rich plasma injection therapies for the management of lateral epicondylitis: A systematic review. SICOT J. 2018;4:11. doi: 10.1051/sicotj/2017062. Epub 2018 Mar 21. PMID 29561260
- [Result] Anitua E, Sanchez M, Nurden AT, Nurden P, Orive G, Andia I. New insights into and novel applications for platelet-rich fibrin therapies. Trends Biotechnol. 2006 May;24(5):227-34. doi: 10.1016/j.tibtech.2006.02.010. Epub 2006 Mar 15. PMID 16540193